CLINICAL TRIAL: NCT00422474
Title: Noninvasive Study of the Time Course of Baroreflex Sensitivity 6-Month After Acute Ischemic Stroke and the Relation of Its Changes With Post Stroke Prognosis
Brief Title: Prognostic Significance of the Baroreflex Sensitivity Changes After Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Dr. Siupak Lee, Far Eastern Memorial Hospital
Other Study IDs: FEMH-95-C-012
Record Dates: First submitted 2007-01-14; First posted 2007-01-17 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Cerebrovascular Accident; Baroreflexes; Autonomic Nervous System Diseases
Keywords: Ischemic stroke; Baroreflex sensitivity; Prognosis; Cardiovascular autonomic regulation
MeSH Terms: conditions — Stroke; Autonomic Nervous System Diseases; Ischemic Stroke

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
After acute stroke, baroreflex sensitivity (BRS) is impaired. This impaired acute stage BRS has been reported to be predictive of worsen outcome years after stroke in general. However, it is not very clear if the impaired acute stroke BRS would actually persist months after the acute stage. It is also not clear that such change, if any, would correlate with the functional outcome or prognosis after stroke.

The trial is to investigate the longitudinal time course of BRS after ischemic stroke up to the 6th month post stroke and to see if there is any correlation of the changes in BRS with the functional outcome parameters using NIHSS and mRS scores throughout this period.

ELIGIBILITY:
Inclusion Criteria:

* Baroreflex sensitivity can be done within 72 hours of onset of acute ischemic stroke
* 50-80 years old
* Must have either brain CT or brain MRI done

Exclusion Criteria:

* NIHSS score > 10
* Patient could not cooperate
* Unstable vital sign
* Atrial fibrillation
* Transient ischemic attack patient
* Diabetic patient
* Impaired renal function (Cr > 2.26 mg/dl)
* Unstable angina, acute myocardiac infarction, cardiomyopathy patients
* Patient who has known autonomic dysfunction

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Siupak Lee, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan